CLINICAL TRIAL: NCT07280130
Title: Evaluation of Occlusal Adjustment Material Removal on Monolithic Zirconia Blocks: An In Vitro Study
Status: Not yet recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202510051RINA
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Dental Occlusion; Occlusal Wear of Teeth; Fixed Dental Prosthesis
Keywords: occlusal adjustment; Monolithic zirconia; Material removal; Silicon carbide stone; 3D scan registration
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- A.fourth-year dental students: Forty fourth-year dental students who have completed preclinical courses in operative dentistry, complete denture prosthodontics, and fixed prosthodontics (Part I). They have little to no experience in adjusting zirconia.
  Interventions: Procedure: perform material removal on monolithic zirconia
- B.sixth-year interns: Forty sixth-year dental interns. Each participant will be tested twice-once before and once near the end of their clinical training. A questionnaire will also record their prosthodontic clinical experience within the past year.
  Interventions: Procedure: perform material removal on monolithic zirconia
- C.clinicians: Forty licensed clinicians with 0-5 years of post-graduation experience (with practical experience in zirconia adjustment). A questionnaire will also document their clinical experience in prosthodontics.
  Interventions: Procedure: perform material removal on monolithic zirconia

INTERVENTIONS:
Procedure: perform material removal on monolithic zirconia — Each participant will perform 100 strokes along an 8-mm path at a rate of 100 strokes per minute, guided by a metronome on the monolithic zirconia

SUMMARY:
This study aims to improve understanding of the amount of tooth-replacement material removed during a single grinding "stroke" performed in the adjustment of a zirconia crown. Zirconia is a highly durable ceramic material commonly used for dental restorations, and accurate adjustment is essential for achieving proper occlusion. However, existing literature does not provide quantitative data regarding material removal per stroke during chairside adjustment, resulting in reliance on individual clinical experience.

In this study, standardized zirconia specimens will be prepared and assigned to three operator groups: dental students, dental interns, and experienced clinicians. Each participant will perform a controlled number of grinding strokes on the specimens using a commonly used dental grinding stone. Specimens will be scanned before and after grinding using a three-dimensional scanner to precisely quantify material removal.

Hypothesis

The hypotheses of this study are:

Each grinding stroke results in a measurable and relatively consistent amount of zirconia material removal.

Experienced clinicians demonstrate more controlled and predictable material removal per stroke compared with students and interns.

DETAILED DESCRIPTION:
Clinical occlusal adjustment requires precision within tens of micrometers; however, current literature lacks objective data regarding per-stroke material removal during chairside adjustment of monolithic zirconia. As a result, clinical decision-making largely depends on subjective judgment.

Objective

The objective of this study is to quantify material removal per single reciprocating grinding stroke on monolithic zirconia blocks using a silicon carbide grinding stone and to compare performance among operators with different levels of clinical experience.

Methods

Monolithic zirconia specimens (VITA YZ ST; dimensions: 8 × 2 × 15 mm) will be milled, sintered, and embedded into standardized holders. Operators will include 40 fourth-year dental students, 40 sixth-year dental interns, and 40 experienced clinicians. Each participant will perform 100 grinding strokes along an 8-mm linear path at a frequency of 100 strokes per minute, guided by a metronome.

Grinding will be performed using a silicon carbide stone (Dura-Green Stone HP 0031/PC2, SHOFU, Japan) operated at 20,000 rpm. Pre- and post-grinding scans will be obtained using a 3Shape F8 scanner. Scan datasets will be superimposed using feature-based alignment to calculate volumetric loss and thickness reduction, expressed as mm³ per stroke and µm per stroke, respectively.

Statistical Analysis

Mixed-effects models will be applied to evaluate group-by-stroke interactions. Reference intervals for material removal will be established, and results will be translated into a clinically applicable occlusal adjustment guide.

Expected Results

The study is expected to define the magnitude and variability of zirconia material removal per grinding stroke, identify differences in performance between operator experience levels, and highlight areas requiring targeted educational training.

Conclusion

This in vitro investigation will provide the first stroke-level quantitative evidence for monolithic zirconia occlusal adjustment. The findings are expected to enhance the accuracy of clinical decision-making, improve training assessment, and support evidence-based guidelines for zirconia crown adjustment.

ELIGIBILITY:
Inclusion Criteria:

Group A: Forty fourth-year dental students who have completed preclinical courses in operative dentistry, complete denture prosthodontics, and fixed prosthodontics (Part I). They have little to no experience in adjusting zirconia.

Group B: Forty sixth-year dental interns. Each participant will be tested twice-once before and once near the end of their clinical training. A questionnaire will also record their prosthodontic clinical experience within the past year.

Group C: Forty licensed clinicians with 0-5 years of post-graduation experience (with practical experience in zirconia adjustment). A questionnaire will also document their clinical experience in prosthodontics.

Exclusion Criteria:

* Acute upper-limb/hand injuries or postoperative recovery within the past 3 months that may affect grip strength or fine motor control.
* Neuromuscular disorders or tremor/postural control impairments (e.g., essential tremor, peripheral neuropathy, moderate to severe carpal tunnel syndrome) that prevent stable operation.
* Uncorrected or inadequately corrected vision that does not meet the requirements for close-range tasks (e.g., inability to clearly see fine markings at a distance of 30-40 cm even with correction).
* Inability to follow the metronome rhythm (100 beats per minute).

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of 120 participants from three levels of dental training and early clinical practice, recruited from a dental school and affiliated clinical institutions. The sample includes:
  1. Fourth-year dental students
  2. Sixth-year dental interns
  3. Clinicians with 0-5 years of post-graduation experience
  Participants are generally healthy adults capable of performing fine motor tasks required for dental procedures. Exclusion criteria include acute hand/upper-limb injuries, neuromuscular disorders, uncorrected poor vision, and inability to follow a metronome rhythm.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The amount of material removal per stroke | about 12 months
  Amount of Zirconia Material Removed per Grinding Stroke(um/stroke)
  * Mean thickness of material removed per stroke
  * Median thickness of material removed per stroke

SECONDARY OUTCOMES:
Change in Material Removal Rate Between Grinding Phases | approximately 12 months
  Difference in mean zirconia material removal per stroke between early grinding phase (strokes 1-50) and late grinding phase (strokes 51-100)
  Unit of Measure: μm/stroke (difference between phases)
Percentile Distribution of Zirconia Material Removal by Operator Experience Level | approximately 12 months
  Percentile distribution (e.g., 25th, 50th, 75th percentiles) of zirconia material removal per grinding stroke within each operator experience group
  Unit of Measure: percentile values

CONTACTS AND LOCATIONS:
Overall Officials: Yihao Lan, DDS, MSD, Study Director — National Taiwan University Hospital

IPD SHARING:
Plan to Share IPD: Undecided
If other research teams conduct similar experiments, we may consider releasing the relevant study data in a de-identified format.